CLINICAL TRIAL: NCT02149238
Title: Acute Study to Investigate the Interaction of Cocoa Methylxanthines With Cocoa Flavanol Related Vascular Effects
Brief Title: Interaction of Cocoa Methylxanthines With Cocoa Flavanol Related Vascular Effects
Acronym: New Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: New Drink
Record Dates: First submitted 2014-05-22; First posted 2014-05-29 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Diseases
Keywords: flavanols; cardiovascular effects; nutrition-nutrition interaction
MeSH Terms: conditions — Cardiovascular Diseases | interventions — methylxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- flavanol rich drink intervention (Active Comparator): flavanol rich drink
  Interventions: Dietary Supplement: flavanol
- methylxanthine rich drink intervention (Active Comparator): methylxanthine rich drink
  Interventions: Dietary Supplement: methylxanthine
- flavanol + methylxanthine rich drink intervention (Active Comparator): flavanol + methylxanthine rich drink
  Interventions: Dietary Supplement: flavanol + methylxanthine

INTERVENTIONS:
Dietary Supplement: flavanol
  Arms: flavanol rich drink intervention
Dietary Supplement: methylxanthine
  Arms: methylxanthine rich drink intervention
Dietary Supplement: flavanol + methylxanthine
  Arms: flavanol + methylxanthine rich drink intervention

SUMMARY:
Epidemiological studies suggest that certain foods rich in flavanols, including cocoa products, red wine, and tea, are associated with decreased cardiovascular mortality and morbidity. Dietary interventional studies have corroborated this finding and showed that flavanols can acutely and after sustained ingestion improve surrogate markers of cardiovascular risk including endothelial function. Endothelial dysfunction is the key event in the development and progression of cardiovascular disease. Aging is the major non-modifiable cardiovascular risk factor associated with progressive decline in endothelial function, vascular stiffening and increase in blood pressure.

However, in addition to flavanols, other potentially bioactive compounds are present in cocoa, in particular methylxanthines. Little is known about the vascular effects of cocoa methylxanthines, i.e. mainly theobromine, in particular when consumed together with flavanols in cocoa products. The aim of the study is to characterize the nutrient-nutrient interaction between cocoa flavanols and cocoa methylxanthines.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* >18 years

Exclusion Criteria:

* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* CRP > 1 mg/dl
* malignant disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 2 hours
  Flow mediated dilatation (FMD)
Plasma flavanol metabolites | 2 hours
  Measured by HPLC

SECONDARY OUTCOMES:
Pulse wave velocity | 2 hours
  Measured by SphygmoCor
Ambulatory blood pressure | 2 hours
  automatical measurements
Circulation angiogenetic cells | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Sansone R, Ottaviani JI, Rodriguez-Mateos A, Heinen Y, Noske D, Spencer JP, Crozier A, Merx MW, Kelm M, Schroeter H, Heiss C. Methylxanthines enhance the effects of cocoa flavanols on cardiovascular function: randomized, double-masked controlled studies. Am J Clin Nutr. 2017 Feb;105(2):352-360. doi: 10.3945/ajcn.116.140046. Epub 2016 Dec 21. PMID 28003203